CLINICAL TRIAL: NCT04758091
Title: The Effect of Tourniquet Application on Optic Nerve Sheath Diameter and Cerebral Oxygenation During Lower Extremity Surgery
Brief Title: Effect of Tourniquet Application on Optic Nerve Sheath Diameter
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Bahar Say, principal investigator, Zonguldak Bulent Ecevit University
Other Study IDs: 2019-58-03/04
Record Dates: First submitted 2021-02-08; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Intracranial Pressure Increase
Keywords: Optic Nerve Sheath Diameter; Tourniquet; Cerebral Oxygenation
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study to investigate the effect of tourniquet application on optic nerve sheath diameter (ONSD) and cerebral oxygenation during lower extremity surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II risk group over the age of 18
* Operation planned under general anesthesia
* Lower extremity surgery with a tourniquet
* Agreeing to volunteer for research with an informed consent form

Exclusion Criteria:

* Emergency surgical procedures
* neurological disease, carotid disease
* Previous intracranial or ocular surgery
* Neurological symptoms
* cerebral edema, high IntraCranial Pressure
* Presence of glaucoma
* Body mass index (BMI)> 35
* Uncontrolled hypertension
* Diabetic retinopathy
* anemia
* coronary artery disease
* peripheral artery disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: lower extremity surgery with tourniquet
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
optic nerve diameter | during the surgery
  measuring the change in optic nerve diameter
regional cerebral oxgenation | during the surgery
  measurement rSo2 by Near Infrared spectroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University Medicine Faculty, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No